CLINICAL TRIAL: NCT05673707
Title: The Effect of Thyromental Height and Other Difficult Airway Evaluation Parameters on Laryngeal Mask Placement Success Rate in Elderly Patients
Brief Title: The Effect of Thyromental Height and Other Difficult Airway Evaluation Parameters
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Savas Altinsoy, Associate Prof, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: LMA
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Airway Complication of Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Thyromental Height — its measure between thyroid and mentum

SUMMARY:
Many changes occur in the body with age. There are difficulties in endotracheal intubation and the placement of supraglottic airway devices (LMA) in elderly patients due to changes in the tooth and facial structure, and a decrease in temporomandibular joint and neck movements. In the literature, there are studies on the relationship between thyromental height measurement and endotracheal intubation difficulty, but there is no study on the relationship between thyromental height measurement and laryngeal mask placement difficulty.

DETAILED DESCRIPTION:
Age, gender, height, body weight, body mass index, type of operation, and Mallampati score are recorded in the preoperative evaluations of all patients. For anthropometric measurements, thyromental height, thyromental distance, sterno-mental distance, neck circumference, and mouth opening are measured. After the laryngeal mask is placed after the induction of anesthesia, the location of the LMA is checked with the FOB (fiberoptic bronchoscopy). Ease of insertion was subjectively assessed using a grading score of 1-4 (1, no resistance; 2, mild resistance; 3, moderate resistance; 4, inability to insert the device) by the attending anesthesiologist who inserted the device. After successful placement of the device, the adjustable pressure limiting (APL) valve is adjusted to 30 cm H2O at 3L/minute fresh gas flow, and the airway pressure and leakage amount are measured.

ELIGIBILITY:
Inclusion Criteria:

* over 65 years old
* elective operation
* using laryngeal mask device

Exclusion Criteria:

* younger than 65 years old
* urgent or emergency operation
* morbidity obese
* contraindications of all laryngeal mask devices using

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: all patients between 65-90 years old who had urological procedure
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
laryngeal mask placement success | during insertion
  The correlation between preoperative thyromental height measurement and laryngeal mask placement success

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Reanimation, University of Health Sciences, Diskapi Yıldırım Beyazit Training and Research Hospital, Ankara, Turkey (Türkiye)